CLINICAL TRIAL: NCT01091701
Title: A Randomized, Double Blind, Multicentric, Placebo Controlled, Single Dose, Phase -I/ II Study Assessing The Safety And Efficacy Of Intravenous Ex Vivo Cultured Adult Allogenic Mesenchymal Stem Cells In Patients With Ischemic Cerebral Stroke
Brief Title: Ex Vivo Cultured Adult Allogenic MSCs in Ischemic Cerebral Stroke
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Collaborators: Stempeutics Research Malaysia SDN BHD (Unknown)
Responsible Party: Dr Anjan K Das, Stempeutics Research Malaysia SDN BHD
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRM/CS/09-10/001
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2011-06

CONDITIONS: Stroke
Keywords: Ischemic Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ex vivo cultured adult allogenic MSCs (Experimental)
  Interventions: Biological: Ex vivo cultured adult allogenic MSCs
- Plasmalyte-A (Placebo Comparator)
  Interventions: Other: Plasmalyte-A

INTERVENTIONS:
Biological: Ex vivo cultured adult allogenic MSCs — Single IV dose of allogenic MSCs
  Arms: Ex vivo cultured adult allogenic MSCs
Other: Plasmalyte-A — Single IV dose of Plasmalyte-A
  Arms: Plasmalyte-A

SUMMARY:
This study will evaluate the safety and efficacy of intravenous ex vivo cultured adult allogenic mesenchymal stem cells in patients with ischemic cerebral stroke. Patient will be given single intravenous dose of allogenic mesenchymal stem cells 2 million cells/Kg body weight or placebo within 10 days of stroke. Patients will be followed up till 12 months. Safety will be evaluated by type, number and proportion of patients with adverse events. Efficacy will be evaluated by clinical parameters and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years old
* MRS equal to or less than 4.
* Full functional independence before present stroke.
* Patients will be included within the time frame of 10 days after an acute cerebral ischemic episode. This time period refers to the date of dosing.
* Neuro-imaging examination showing ischemic cerebral infarct.
* CT or MRI brain scanning has reliably excluded both intracranial haemorrhage and structural brain lesions which can mimic stroke (e.g. cerebral tumour)
* Stroke symptoms are to be present for at least 30 minutes and have not improved before treatment. Symptoms must be distinguishable from an episode of generalized ischemia (i.e. syncope), seizure, or migraine disorder. Patients should have motor weakness following the acute cerebral ischemic episode.
* Able to comply with study procedures for the entire length of the study

Exclusion Criteria:

* Haematological causes of stroke
* Evidence of intracranial haemorrhage (ICH) on the CT-scan.
* Severe stroke as assessed clinically (e.g. MRS>4).
* Subjects who are unlikely to complete the infusion of investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation, intra cranial surgery or radiological evidence of previous cerebral stroke with clinical manifestation.
* History of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Size and location of the cerebral infarct cannot be determined.
* Comatose / clinically unstable
* Serious, pre-existing medical conditions such as bleeding disorders (eg. leukopenia, thrombocytopenia) septicemia, TB, hepatic dysfunction (> 2.5 times the ULN of hepatic function tests) and renal dysfunction (Serum creatinine > 2 mg/dl).
* Disease or impairment that precludes adequate neurological exam
* Hypo- or hyperglycaemia sufficient to account for the neurological symptoms; the patient should be excluded if their blood glucose is < 3.0 or > 20.0mmol/L.
* The patient is female and of childbearing potential (unless it is certain that pregnancy is not possible) or breast feeding.
* Patient is likely to be unavailable for follow-up e.g. no fixed home address
* Patients with evidence of life threatening infection or life threatening illness (e.g. advanced cancer) or having tested positive for HIV, Hepatitis B, Hepatitis C and VDRL
* Patient was already dependent in activities of daily living before the present acute stroke
* Patients who have been included in any other clinical trial within the previous month
* History of neoplasia or other comorbidity that could impact patient's short-term survival
* Previous or concomitant treatment with immune modulators or experimental drugs 60 days prior to study enrolment
* Any condition that in the judgment of the investigator would place the patient under undue risk
* Sustained systolic BP >220 mmHg, or <80mmHg, or diastolic BP > 140mmHg or <50 mmHg.
* Patients contraindicated for MRI examination.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The type of AE(s), number of AE(s) and proportion of patients with AE(s). | 12 Months
Improvement of neurological recovery as assessed by NIH Stroke Scale (NIHSS). | 12 Months

SECONDARY OUTCOMES:
Improvement of the Functional recovery - assessed by Barthel's Index for activities of daily living. | 12 Months
Improvement of Global outcome as assessed by the Modified Rankin Scale | 12 Months
MRI Parameters - Change in infarct size T2 - weighted images and blood flow in infarct area as evaluated by Diffusion Weighted Index | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abdul Syukur Abdullah, MD, Principal Investigator — Hospital Sultanah Bahiyah Consultant Physician, Medical Department, Km 6 Jalan Langgar, 5460 Alor Setar, Kedah; Dr Irene Looi, MD, Principal Investigator — Hospital Seberang jaya Jalan Tun Hussein Onn 13700 Prai, Pulau Pinang; Dr Uduman Ali Mohamed Yousuf, MD, Principal Investigator — Hospital Melaka Consultant Neurologist, Neurology Clinic, Medical Department, Jalan Mufti Haji Khalil, 75400 Melaka; Dr Dato K Chandran, MD, Principal Investigator — Hospital Raja Permaisuri Bainun Consultant Physician, Jalan Hospital, 30990,Ipoh, Perak; Dr Chuah Siew Kee, MD, Principal Investigator — Hospital Sungai Buloh Consultant Physician, Department of Medicine, Jalan Hospital, 47000 Sungai Buloh, Selangor; Dr Yau Weng Keong, MD, Principal Investigator — Hospital Kuala Lumpur Consultant Physian and Geriatrician, Jalan Pahang, 50586 Kuala Lumpur
Locations (6):
- Malaysia (6):
  - Hospital Raja Permaisuri Bainun, Jalan Hospital, 30990,, Ipoh, Perak
  - Hospital Kuala Lumpur, Jalan Pahang, 50586, Kuala Lumpur
  - Hospital Melaka, Jalan Mufti Haji Khalil, 75400, Melaka
  - Hospital Seberang jaya Jalan Tun Hussein Onn, 13700, Perai, Pulau Pinang
  - Hospital Sungai Buloh, Jalan Hospital, 47000, Sungai Buloh, Selangor
  - Hospital Sultanah Bahiyah, Km 6 Jalan Langgar, 5460 Alor Setar, Kedah